CLINICAL TRIAL: NCT05948631
Title: MISC-IPV: a Community-Based Intervention for Children Traumatized by Intimate Partner Violence
Acronym: MISC-IPV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Houston (Other)
Collaborators: Texas Women's University (Unknown)
Responsible Party: Principal Investigator, Carla Sharp, John and Rebecca Moores Professor and Associate Dean, University of Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00001728
Record Dates: First submitted 2023-06-16; First posted 2023-07-17 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: MISC Intervention; Treatment As Usual
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MISC (Experimental): Mediational Intervention for Sensitizing Caregivers (MISC): a program for mother and children where mothers become sensitized to the impact of their behavior on their children with the aim of improving quality caregiving and child outcomes.
  Interventions: Behavioral: MISC intervention
- Treatment as Usual (Active Comparator): Treatment as Usual in the rehousing program. Mothers receive support in a domestic violence rehousing program to find work and housing.
  Interventions: Behavioral: Treatment as Usual (TAU)

INTERVENTIONS:
Behavioral: MISC intervention — MISC is a semi-structured, participatory caregiver intervention following these steps: (1) Identify the mother's personal and cultural characteristics, which include a respectful discussion around the mother's child-rearing views, objectives, needs and expectations. (2) Create a baseline through videotaped interactions. (3) Create caregivers' personal interaction profile on the basis of videotaped interaction. The caseworker builds on the initial videotaped interaction and uses subsequent bi-weekly videotaped interactions to give feedback to mothers on the frequency of mediational behaviors thereby quantifying the quality of mother-child interactions. Interactional characteristics are jointly identified and conceptualized according to MISC principles. The mother learns to understand both her own and the child's behavior within a meaningful framework, enhancing reflection of caregiving practices. (4) In-service training (once a month). (5) Re-evaluate training efficacy.
  Arms: MISC
Behavioral: Treatment as Usual (TAU) — TAU consists of supportive services including trauma informed, client-centered, and strength-based case management and advocacy. All services are focused on the mother and do not include any child-focused intervention. Instead, staff provide in-home intensive case management services to assess and provide safety planning, assess other social service needs, link abused mothers to community resources, and assist clients in rehousing. TAU direct contact with the mother consists of bi-weekly contact, which matches the contact frequency for the intervention group. However, MISC mothers will be receiving TAU+MISC-IPV (2 hours bi-weekly contact) compared with TAU only (30 minutes biweekly contact).
  Arms: Treatment as Usual

SUMMARY:
This study adapts and evaluates preliminary outcomes of the Mediational Intervention for Sensitizing Caregivers (MISC) for women and children of color who have survived domestic violence.

DETAILED DESCRIPTION:
The investigators propose that the adverse effects of Intimate Partner Violence (IPV) trauma on children can be interrupted through an intervention that enhances maternal caregiving capacity delivered by paraprofessional caseworkers. The objective of this application is to adapt an established caregiver intervention program, Mediational Intervention for Sensitizing Caregivers (MISC), for the IPV context (thereafter named MISC-IPV). Guided by an evidence-based framework for adapting caregiver-child training programs, the investigators take a three-phase approach (Adapt, Process Evaluation, Outcome/Mediator Evaluation) with the central hypothesis that acceptability and feasibility of MISC-IPV will be demonstrated and that MISC-IPV will show positive preliminary outcomes through the mechanism of enhanced maternal caregiving. In acknowledgement of significant health disparities faced by IPV-affected African American women, the investigators will conduct our research with African American women and their children. Successful completion of the project will result in a scalable community-based approach to IPV exposure that may provide a model for future integration of child-focused work into existing woman-focused IPV programs.

ELIGIBILITY:
Mother inclusion criteria:

1. Enrolled in Harris County Domestic Violence rehousing program
2. Fluency in English

Mother exclusion criteria:

1. Active suicidality
2. Intellectual disability
3. Active psychotic disorder

Child inclusion criteria:

1. Exposure to domestic violence
2. 7-11 years old in a family

Child exclusion criteria:

1. Intelligence quotient below 75,
2. Active psychosis
3. Severe autism
4. Below age 7 or above age 11

Ages: 7 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2023-02-14 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Mental health problems | Baseline, six, 12, and 18 months.
  The primary outcome measure is change in mental health outcomes as assessed through by the Strengths and Difficulties Questionnaire (SDQ). The SDQ total score indexes the overall level of mental health problems a child is experiencing with a minimum score of 0 and a maximum score of 60. A higher the score indicates higher the levels of mental health problems.
Sensitive caregiving | Baseline, six, 12, and 18 months.
  Change in sensitive caregiving is a primary outcome that will be assessed with an observational tool named the Observing Mediational Interaction (OMI) tool. The measure codes the frequency of caregiving behaviors that are sensitive to the child's needs. It has a minimum of 0, but has no maximum as any frequency of behaviors may be observed. A higher score indicates more sensitive caregiving.

CONTACTS AND LOCATIONS:
Overall Officials: Carla Sharp, Principal Investigator — csharp2@uh.edu
Locations (1):
- University of Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided